CLINICAL TRIAL: NCT05338762
Title: Clinical Agreement Study of 'TekiTrustTM SARS-CoV-2 Neutralizing Antibody Detection ELISA Kit' and 'TekiTrustTM SARS-CoV-2 Neutralizing Antibody Detection Rapid Test'
Brief Title: TekiTrust Tests to Determine the Level of SARS-COV-2/COVID-19 Neutralizing Antibodies in the Blood
Status: Completed | Type: Observational
Sponsor: MiCo BioMed Co., Ltd. (Industry)
Collaborators: Syntactx (Network)
Responsible Party: Sponsor
Other Study IDs: MIC-US-2021-001
Record Dates: First submitted 2021-06-02; First posted 2022-04-21 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: SARS-CoV2 Infection
Keywords: Antibodies, Neutralizing; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Current COVID-19 symptoms or SARS-CoV-2 in the last 30 days with a positive RT-PCR test: 75 subjects will be enrolled who were diagnosed as SARS-CoV-2 with a positive RT-PCR nasal pharangeal test or are suspected of having a COVID-19 infection with symptom onset in the last 30 days. (Symptom onset 0-30 days)
  This group of subjects will receive:
  1. a fingerstick blood sample for a rapid test neutralizing antibody test to be done in the office with the TekiTrust SARS-CoV-2 Neutralizing Antibody Detection Rapid Test
  2. a blood draw which will be sent to the lab for neutralizing antibody testing with the TekiTrust SARS-CoV-2 Nuetralizing Antibody Detection ELISA Kit and the standard Plaque Reduction Neutralization Test (PRNT)
  3. a nasal-pharangeal RT-PCR test
- Diagnosed with SARS-CoV-2 (COVID-19) in the past 3 months with a positive RT-PCR test: 30 subjects will be enrolled who have been diagnosed with COVID-19 in the past 3 months and had a prior positive RT-PCR nasal pharangeal test. (Symptom onsent 31-90 days)
  This group of subjects will receive:
  1. a fingerstick blood sample for a rapid test neutralizing antibody test to be done in the office with the TekiTrust SARS-CoV-2 Neutralizing Antibody Detection Rapid Test
  2. a blood draw which will be sent to the lab for neutralizing antibody testing with the TekiTrust SARS-CoV-2 Nuetralizing Antibody Detection ELISA Kit and the standard Plaque Reduction Neutralization Test (PRNT)

SUMMARY:
The purpose of this study is to determine if the TekiTrust Enzyme-Linked Immunosorbent Assay (ELISA) Kit and TekiTrust Rapid Test can accurately determine the amount of antibodies to fight the COVID-19 virus in sampled blood compared to the standard Plaque Reduction Neutralization Test (PRNT) test.

When a person has COVID-19 they develop antibodies to the virus which are contained in their blood stream. After a certain period, the number of antibodies to fight (neutralize) the virus begin to decrease. One common way to measure the amount of antibodies in the blood is to use a test called the PRNT. The focus of this study is to compare the ability of the TekiTrust ELISA Kit and the TekiTrust Rapid Test with the PRNT to determine if these tests can measure the antibodies equally well.

DETAILED DESCRIPTION:
Participants who have been previously diagnosed with COVID-19 within the past 3 months through any FDA emergency use approved (EUA) assay test will eligible for inclusion in the study. A blood and fingerstick sample will be obtained from the participant and for subjects with a positive test and symptom onset of less than 30 days a repeat RT-PCR nasal pharyngeal swab sample will be taken. The fingerstick sample will be used onsite by qualified site staff to test the TekiTrust SARS-CoV-2 Neutralizing Antibody Detection Rapid Test. These results will be compared to the whole blood sample sent to the lab which will be analysed for SARS CoV-2 neutralizing antibodies using the TekiTrust SARS-CoV-2 Neutralizing Antibody Detection ELISA Kit and the comparator Plaque Reduction Neutralization Test (PRNT) test.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Able and willing to provide written informed consent
3. Previously diagnosed as SARS-CoV-2 positive by any FDA EUA approved assay with a symptom onset date within the previous 30 days and who are willing to provide a nasopharyngeal swab for RT-PCR testing
4. Suspected of previous SARS-CoV-2 infection and willing to provide a nasopharyngeal swab for RT-PCR testing
5. Previously diagnosed as SARS-CoV-2 positive by a FDA EUA approved RT-PCR assay with a symptom onset date greater than 30 days and a known date of PCR sample collection and symptom severity

Exclusion Criteria:

1. Any significant medical, psychological, or social condition which in the opinion of the investigator may preclude the subject from participating in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Participants who have been previously diagnosed with SARS-CoV-2 through any FDA Emergency Use Authorization (EUA) approved assays with symptom onset within the previous 30 days or who are suspected of SARS-CoV-2 infection and are tested with FDA EUA approved RT-PCR.
  2. Participants who have previously been diagnosed with SARS-CoV-2 through an FDA EUA approved RT-PCR assay with recorded symptom onset date more than 30 days, from date of PCR sample collection.
Sampling Method: Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Clinical agreement between TekiTrust SARS-CoV-2 Neutralizing Antibody ELISA Kit and Rapid Detection test and the comparator PRNT assay. | Day one
  1. PPA (Sensitivity) between ≥87% with a lower bound of the 95% confidence interval greater than 74.4%
  2. NPA (Specificity) ≥ 93% with a lower bound of the 95% confidence interval greater than 87.8%

SECONDARY OUTCOMES:
Safety endpoint: adverse events | Single study visit
  Number of adverse events related to blood sample testing in tested participants.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Hahn, PhD, Study Director — MiCo BioMed
Locations (5):
- United States (5):
  - Mississippi State University, Starkville, Mississippi
  - Joy Internal Medicine, Englewood Cliffs, New Jersey
  - WellNow Urgent Care, Cincinnati, Ohio
  - WellNow Urgent Care, Columbus, Ohio
  - WellNow Urgent Care, Dayton, Ohio

IPD SHARING:
Plan to Share IPD: No